CLINICAL TRIAL: NCT04209062
Title: Validation of a High-Quality Low-Cost Open-Source Electrocardiograph (ECG)
Brief Title: Validation of a High-Quality Low-Cost Open-Source Electrocardiograph
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Tarek Loubani, MD, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 112365
Record Dates: First submitted 2018-08-13; First posted 2019-12-23 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Open Access; Medical Devices; Low Cost; Electrocardiograph
Keywords: Open Access; Medical Devices; Low Cost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study device (Experimental)
  Interventions: Device: Medical device validation
- Control device (Active Comparator)
  Interventions: Device: Medical device validation

INTERVENTIONS:
Device: Medical device validation — The medical devices will both record electrical signals for comparison

SUMMARY:
The high price of electrocardiograph (ECG) devices - with most hospital-grade devices costing thousands of dollars - is one of the barriers to access of this vital technology. There is a shortage of ECG devices in underserved areas and the devices available on the market currently are not adequate to solve this problem. Our solution is a low-cost high-quality open-access ECG device. This study intends to validate the study ECG device in human patients by demonstrating equivalence between the study ECG device and a gold standard device.

ELIGIBILITY:
Inclusion Criteria:

- All study participants must be able to provide written informed consent prior to study procedure. This study has 2 Phases.

Phase 1:

* Healthy
* > 18 years of age

Phase 2:

* > 18 years of age
* non critical patients presenting to the emergency department (Victoria Hospital and University Hospital) with cardiac complaint

Exclusion Criteria:

* < 18 years old
* Unable to consent

Phase 1:

* > 70 years of age
* Previous history of cardiac disease (e.g., atrial fibrillation, myocardial infarction, congestive heart failure)
* current status of non-sinus heart rhythm

Phase 2:

- Critical patients in the ED where consent would inappropriately delay investigations or treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Equivalence of Electrical Signals between 3D printed ECG device and Gold Standard ECG | 60 seconds
  Comparing electrical signals from ECG electrodes with tested device and gold standard device by collecting the following data from both devices: rate, QR interval, PR interval, QT interval, and rhythm.

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No